CLINICAL TRIAL: NCT02557997
Title: Effects of Dolutegravir Based Regimen on HIV-1 Reservoir and Immune Activation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6074
Record Dates: First submitted 2015-09-14; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: HIV-1 Infection
Keywords: HIV reservoir; HIV-1 DNA; Immune activation; Monocyte function; Activation biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ART-naive (primary infection): ART-naive (primary infection) HIV infected adults
  Interventions: Other: Blood tube bottom analyses
- ART-naïve (chronic infection): ART-naïve (chronic infection) HIV infected adults
  Interventions: Other: Blood tube bottom analyses
- ART-controlled: ART-controlled HIV infected adults
  Interventions: Other: Blood tube bottom analyses
- ART-failing: ART-failing HIV infected adults
  Interventions: Other: Blood tube bottom analyses

INTERVENTIONS:
Other: Blood tube bottom analyses

SUMMARY:
We aim at comparing markers of HIV reservoir, monocyte function and immune activation between antiretroviral therapy (ART)-naïve (chronic infection or primary infection), ART-controlled or ART-failing HIV infected adults initiating a dolutegravir (DTG)-based regimen. The investigators' purpose is to measure cell associated HIV-1 DNA, monocyte function [soluble CD14 (sCD14), soluble CD163 (sCD163)], and immune activation [neopterine, interleukin-6 (IL-6) and high-sensitivity C-reactive protein (hsCRP)] biomarkers at different time points between baseline and week 48 post DTG-based regimen initiation in each group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from de 18 to 80 years
* Patient starting a DTG-regimen
* Patients agreeing to use methods of birthcontrol while on the study and during the 6 weeks after stopping DTG treatment
* Signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* HBV or HCV coinfection
* Participation in another clinical drug or device trial where the last dose of drug was within the past 30 days or an investigational medical device is currently implanted
* Documented resistance to DTG
* Allergy or intolerance to the study drugs or their components or drugs of their class
* Any acute or verified Grade 4 laboratory abnormality (with the exception of Grade 4 lipids) at Screening.
* Coadministration with Dofelitide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting an HIV Infection care center at a university hospital will be selected
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Proviral HIV-1 DNA at Week 48 | Baseline and 48 weeks post DTG-based regimen initiation

SECONDARY OUTCOMES:
Quantification of biomarkers of immune activation | Baseline, 24 and 48 weeks post DTG-based regimen initiation
  Soluble CD14 (sCD14), soluble CD163 (sCD163), neopterine, interleukin-6 (IL-6), high-sensitivity C-reactive protein (hsCRP)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg - Trait d'Union, Strasbourg, France

REFERENCES:
- [Derived] Gantner P, Barnig C, Partisani M, Lee GQ, Beck-Wirth G, Faller JP, Martinot M, Mosheni-Zadeh M, Cheneau C, Batard ML, Fischer P, Fuchs A, Uring-Lambert B, Bahram S, Rey D, Fafi-Kremer S. Distribution and reduction magnitude of HIV-DNA burden in CD4+ T cell subsets depend on art initiation timing. AIDS. 2018 Apr 24;32(7):921-926. doi: 10.1097/QAD.0000000000001770. PMID 29424775
- [Derived] Gantner P, Lee GQ, Rey D, Mesplede T, Partisani M, Cheneau C, Beck-Wirth G, Faller JP, Mohseni-Zadeh M, Martinot M, Wainberg MA, Fafi-Kremer S. Dolutegravir reshapes the genetic diversity of HIV-1 reservoirs. J Antimicrob Chemother. 2018 Apr 1;73(4):1045-1053. doi: 10.1093/jac/dkx475. PMID 29244129